CLINICAL TRIAL: NCT02314052
Title: Phase 1b/2, Multicenter, Dose Escalation Trial to Determine the Safety, Tolerance, Maximum Tolerated Dose and Recommended Phase 2 Dose of DCR-MYC, a Lipid Nanoparticle (LNP)-Formulated Small Inhibitory RNA (siRNA) Oligonucleotide Targeting MYC, in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Phase Ib/2, Multicenter, Dose Escalation Study of DCR-MYC in Patients With Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCR-MYC-102
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCR-MYC (Experimental): Patient groups (cohorts) will receive a single dose level of DCR-MYC; the dose level of DCR-MYC will be increased in subsequent cohorts
  Interventions: Drug: DCR-MYC

INTERVENTIONS:
Drug: DCR-MYC — Dosing: 2 hour IV infusion on Day 1 and 8 of each 21 day cycle.
  Starting dose: 0.125mg/kg/dose
  Number of cycles: until progression or unacceptable toxicity develops.
  PHASE 1b Dose escalation: 50% or 25% increase in subsequent cohorts depending upon toxicity until maximum tolerated dose (MTD) is identified.
  PHASE 2 Cohort expansion at the MTD: Additional patients to be treated at the highest dose tolerated to assess efficacy and further assess safety

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the investigational anticancer drug DCR-MYC. DCR-MYC is a novel synthetic double-stranded RNA in a stable lipid particle suspension that targets the oncogene MYC. MYC oncogene activation is important to the growth of many hematologic and solid tumor malignancies. In this study the Sponsor proposes to study DCR-MYC and its ability to inhibit MYC and thereby inhibit cancer cell growth.

DETAILED DESCRIPTION:
In this second study in humans, DCR-MYC will be administered by 2 hour intravenous (IV) infusion, once weekly for 2 weeks followed by a rest week (3 weeks = 1 cycle), to patients with hepatocellular carcinoma who are either sorafenib-refractory, sorafenib-intolerant despite dose reduction and best supportive care, or for whom neither sorafenib nor other suitable therapy is available. During the Phase 1b portion of the study, the highest safe dose of DCR-MYC that can be administered will be identified. In addition, the pharmacokinetic (PK) profile, potential pharmacodynamic (PD) effects, as well as the preliminary antitumor activity of DCR-MYC will be evaluated. During the Phase 2 portion of the study, up to 30 patients will be treated at the MTD identified in Phase 1b in order to further evaluate safety and tolerability, as well as assess the antitumor activity, of DCR-MYC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, > 18 years of age (in Singapore > 21 years or > 18 years with consent of guardian).
2. Patients with documented (histologically- or cytologically-proven) HCC, with at least 1 measureable lesion > 10 mm (excluding bone metastases). If the measurable lesion(s) is in the liver, it either should not have been treated previously with loco-regional therapy, or there must be demonstrated progression of the lesion following previous loco-regional therapy.
3. Patients with Barcelona Clinic Liver Cancer (BCLC) stage B or C HCC not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
4. Patients who are either refractory to or intolerant of sorafenib despite dose reduction and best supportive care, or patients who do not have access to sorafenib or other suitable therapy for HCC.
5. Patients with underlying hepatic cirrhosis must have a current cirrhosis status of Child-Pugh Class A (i.e., score of 5-6) without encephalopathy.
6. Phase 1b MTD Biopsy Cohort: Patients with primary or metastatic tumor site(s) considered safely accessible for biopsy and consenting to undergo pre- and post-dosing tumor biopsies.
7. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and an anticipated life expectancy of ≥ 3 months.
8. Patients, both male and female, who are either not of childbearing potential or who agree to use a medically effective method of contraception during the study and for 3 months after the last dose of study drug.
9. Patients with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria (Patients):

1. Women who are pregnant or lactating; women of child-bearing potential (WOCBP), and fertile men with a WOCBP-partner not using and not willing to use a medically effective method of contraception.
2. Patients with known central nervous system (CNS) or leptomeningeal metastases not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
3. Patients with mixed histology cholangiocarcinoma and HCC, or fibrolamellar variant HCC.
4. Patients with any of the following hematologic abnormalities at baseline:

   * Hemoglobin < 8.5 g/dL
   * Absolute neutrophil count < 1,500 per mm3
   * Platelet count < 75,000 per mm
5. Patients with any of the following serum chemistry abnormalities at baseline:

   * Total bilirubin > 1.5 × the upper limit of normal (ULN) for the institution
   * AST or ALT > 5 × the ULN for the institution
   * Serum creatinine > 1.5 × the ULN for the institution
6. Patients with the following coagulation parameter abnormality at baseline:

   * INR > 1.7 × ULN for the institution
7. Patients with:

   * A history of deep vein thrombosis (DVT) or pulmonary embolism (PE), within 6 months prior to first study drug administration; patients receiving systemic anti-coagulation for prophylactic or therapeutic reasons
   * Active uncontrolled bleeding or a known bleeding diathesis
8. Patients with:

   * Esophageal or gastric variceal bleeding within 2 months prior to first study drug administration; patients with a history of variceal bleeding between 2 and 12 months prior to first study drug administration should have undergone adequate treatment and be considered clinically stable in the opinion of the investigator
   * A history of symptomatic ascites requiring paracentesis within the past 3 months or any encephalopathy requiring hospitalization or medication within the past 3 months
   * Portal-caval shunts
9. Patients with a significant cardiovascular disease or condition, including:

   * Congestive heart failure currently requiring therapy
   * Need for antiarrhythmic medical therapy for a ventricular arrhythmia
   * Severe conduction disturbance (i.e., 3rd degree heart block)
   * Angina pectoris requiring therapy
   * Known left ventricular ejection fraction (LVEF) < 50% by MUGA or echocardiogram
   * QTc interval > 450 msec in males, or > 470 msec in females
   * Uncontrolled systemic hypertension (per the Investigator's discretion)
   * Class III or IV cardiovascular disease according to the New York Heart Association (NYHA) Functional Criteria
   * Myocardial infarction within 6 months prior to first study drug administration
10. Patients with a known or suspected hypersensitivity to any of the components of lipid nanoparticle-formulated DCR-MYC; patients with a known sensitivity to cremophor (found with paclitaxel and other formulations).
11. Patients with an estimated daily alcohol intake greater than 80 g/day.
12. Patients having undergone previous organ transplantation (e.g., liver transplantation) requiring immunosuppression; patients on long-term immunosuppressive therapy.
13. Patients with a known history of human immunodeficiency virus (HIV) seropositivity.
14. Patients with any other serious/active/uncontrolled infection, with the exception of chronic hepatitis B virus (HBV) or chronic hepatitis C virus (HCV) infection; any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 2 weeks prior to first study drug administration.
15. Patients with inadequate recovery from an acute toxicity associated with any prior antineoplastic therapy.
16. Patients with inadequate recovery from any previous surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to first study drug administration.
17. Patients with an active second malignancy or history of another malignancy within the last 3 years, with the exception of:

    * Treated, non-melanoma skin cancers
    * Treated CIS of the breast or cervix
    * Controlled, superficial carcinoma of the bladder
    * T1a or b carcinoma of the prostate treated according to local standard of care, with prostate specific antigen (PSA) within normal limits (wnl)
18. Patients with any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug.
19. Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study-related evaluations.
20. Patients with the inability or with foreseeable incapacity, in the opinion of the Investigator, to comply with the protocol requirements, including the ability to attend all visits and undergo all assessments.

Exclusion Criteria (Treatments):

1. Phase 1b: Greater than 3 prior systemic anti-cancer chemotherapies or targeted agents for HCC; prior loco-regional treatment, including transcatheter arterial chemo-embolization (TACE), is allowed.
2. Phase 2: greater than 1 prior systemic anti-cancer chemotherapy or targeted agent for HCC; prior loco-regional treatment, including TACE, is allowed.
3. Sorafenib therapy within 2 weeks prior to first study drug administration and during study.
4. Any other antineoplastic agent (standard or experimental) within 4 weeks; monoclonal antibody therapy, nitrosoureas, and nitrogen mustard within 6 weeks prior to first study drug administration and during study.
5. Loco-regional therapy including TACE or radioembolization within 6 weeks prior to first study drug administration and during study.
6. Radiotherapy within 4 weeks prior to first study drug administration and during study.
7. Therapy with sofosbuvir for HCV within 6 weeks prior to first study drug administration and during study.
8. Herbal preparations, or related non-prescription preparations/supplements containing herbal ingredients, aimed at treating the underlying malignancy within 2 weeks prior to first study drug administration and during study.
9. Systemic hormonal therapy within 2 weeks prior to first study drug administration and during study.
10. Any other investigational treatments during study. This includes participation in any medical device or therapeutic intervention clinical trial.
11. Prophylactic use of hematopoietic growth factors within 1 week prior to first study drug administration and during Cycle 1 of study; thereafter prophylactic use of growth factors is allowed as clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Singapore (2):
  - National University Hospital of Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: N = 3, received two, 2-hour infusions of 0.125 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined five 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 2: N = 3, received two, 2-hour infusions of 0.2 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined five 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 3: N = 3, received two, 2-hour infusions of 0.3 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined five 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 4: N = 3, received two, 2-hour infusions of 0.45 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined five 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 5: N = 6, received two, 2-hour infusions of 0.68 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined five 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 6: N = 3, received two, 2-hour infusions of 0.85 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined five 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
Period: Cycle One
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 3 | 3 | 3 | 6 | 3
Completed | 3 | 3 | 3 | 2 | 6 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Cycle Two
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 3 | 3 | 2 | 6 | 3
Completed | 3 | 2 | 2 | 1 | 2 | 3
Not Completed | 0 | 1 | 1 | 1 | 4 | 0
Period: Cycle Three
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 2 | 2 | 1 | 2 | 3
Completed | 3 | 2 (1 of 2 completers in cohort 2 (subject 02-005) only completed 1 of 2 infusions during this cycle) | 2 | 1 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cycle Four
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 2 | 2 | 1 | 2 | 3
Completed | 0 | 2 | 1 | 0 | 2 | 0
Not Completed | 3 | 0 | 1 | 1 | 0 | 3
Period: Cycle Five
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 0 | 2 | 1 | 1 (subject missed cycle four but returned for cycle 5) | 2 | 0
Completed | 0 | 0 | 0 | 1 (subject missed cycle four but returned for cycle 5) | 2 | 0
Not Completed | 0 | 2 | 1 | 0 | 0 | 0
Period: Cycles 6 -10.5
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 0 | 0 | 0 | 1 | 2 | 0
Completed | 0 | 0 | 0 | 1 | 2 (Subject 02-014 only completed 1 of 2 doses in cycle 6) | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DCR-MYC: Patient groups (cohorts) will receive a single dose level of DCR-MYC; the dose level of DCR-MYC will be increased in subsequent cohorts
  DCR-MYC: Dosing: 2 hour IV infusion on Day 1 and 8 of each 21 day cycle.
  Starting dose: 0.125mg/kg/dose
  Number of cycles: until progression or unacceptable toxicity develops.
  PHASE 1b Dose escalation: 50% or 25% increase in subsequent cohorts depending upon toxicity until maximum tolerated dose (MTD) is identified.
  PHASE 2 Cohort expansion at the MTD: Additional patients to be treated at the highest dose tolerated to assess efficacy and further assess safety
Arm/Group | DCR-MYC
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 8
  Singapore | 7
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Part A: 3 patient cohorts with 50% dose increase between cohorts until study drug-related dose-limiting toxicity (DLT) during Cycle 1, then expand to 6 patients and move to Part B.
  Part B: 3 to 6 patient cohorts with 25% dose increase between cohorts until > 1 study drug-related DLT, then stop escalation.
  Expand MTD cohort to 12 patients; tumor biopsies to be performed in this Phase 1b MTD Biopsy Cohort (6 patients).
Time Frame: Cycle 1 (3 weeks), longer if DCR-MYC is continued; with 30 days follow-up after last dose
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3
Participants | 3 | 3 | 3 | 3 | 6 | 3

2. Primary Outcome: Phase 2: Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Up to 30 patients in the Phase 2 MTD Expansion Cohort (to be treated at the MTD identified in Phase 1b); further evaluation of safety and tolerability.
Time Frame: Cycle 1 (3 weeks), longer if DCR-MYC is continued; with 30 days follow-up after last dose
Population: N/A - Study terminated prior to Phase 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 2: Preliminary Antitumor Activity
Description: Up to 30 patients in the Phase 2 MTD Expansion Cohort (to be treated at the MTD identified in Phase 1b); evaluation for evidence of objective response or disease stabilization.
Time Frame: After Cycle 2 (6 weeks), then at 6 week intervals if DCR-MYC is continued
Population: N/A - Study terminated prior to phase 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Cmax (ng/mL) - DCR-MYC Levels in Blood (Phase 1b Only): Dosing Day 1 and Day 8
Description: Samples to be collected Week 1 (Day 1, 2, and 4) and Week 2 (Day 8 and 11). A summary of outcome measures reported here are noncompartmental PK parameters (Cmax, dose-normalized Cmax (Cmax_D), Tmax, AUClast, and dose-normalized AUClast (AUClast_D)) for both infusion days (Day 1 and Day 8).
Time Frame: Week 1 Day 1 AND Week 2 Day 8 Cycle PK Sampling Points: 0 min, 1/4 through infusion, 1/2 through infusion, end of infusion, 15 min, 30 min, 1h, 2h, 4h, 6h, 8h, 24h, Day 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3
ng/mL
  Cmax: Day 1 | 2094.3 (1257.8) | 4790.5 (3540.2) | 6195.7 (744.75) | 9807.1 (4094.5) | 19399 (8211.4) | 19829 (3686.2)
  Cmax: Day 8 | 1755.7 (59.47) | 5504.9 (3365.3) | 6628.4 (1155.8) | 13484 (2576.2) | 20711 (13768) | 27067 (9105.1)

5. Secondary Outcome: DCR-MYC Biological Activities (Phase 1b Only)
Description: Collection of blood samples for cytokine measurements (Day 1, 2, and 4). No noteworthy increases were observed across dose groups or time for GM-CSF, IFNα, IFNɣ, or IL-1β. Changes that were observed for the other cytokines were not dose-dependent since they occurred sporadically and primarily in Cohorts 3 (0.3 mg/kg) and 4 (0.45 mg/kg). Pre-dose, 4 hours post-dose, and 24 hour post-dose results for TNF-α, IL-10, IL-6, IL-8, IL-1RA, and MCP-1 are summarized here.
Time Frame: Cycle 1; Week 1
Population: Safety population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3
pg/mL
  TNF-α Pre-dose | 2.3 (1.3) | 1.6 (0) | 4.1 (0.7) | 1.6 (0) | 3.1 (3.0) | 1.6 (0)
  TNF-α 4 hour post-dose | 1.6 (0) | 1.6 (0) | 15.9 (16.6) | 23.1 (34.2) | 1.6 (0) | 1.6 (0)
  TNF-α 24 hour post-dose | 1.6 (0) | 4.1 (0.5) | 4.5 (1.2) | 3.3 (2.9) | 2.4 (1.7) | 3.8 (3.8)
  IL-10 pre-dose | 317.5 (60.9) | 239.4 (83.7) | 741.1 (46.7) | 574.3 (341.0) | 670.2 (369.4) | 599.7 (333.8)
  IL-10 4 hour post | 241.1 (61.3) | 159.6 (104.2) | 933.1 (427.2) | 1316.7 (1617.7) | 527.1 (225.5) | 533.7 (265.6)
  IL-10 24 hour post | 322.5 (152.9) | 424.4 (296.4) | 939.3 (939.3) | 667.7 (362.7) | 541.8 (240.9) | 830.7 (333.3)
  IL-6 pre-dose | 1.6 (0) | 1.6 (0) | 1.6 (0) | 1.6 (0) | 1.6 (0) | 7.9 (10.9)
  IL-6 4 hour post-dose | 1.6 (0) | 1.6 (0) | 38.3 (51.9) | 133.7 (228.7) | 1.6 (0) | 4.7 (5.3)
  IL-6 24 hour post-dose | 2.2 (1.0) | 1.6 (0) | 6.3 (6.6) | 1.6 (0) | 3.8 (3.8) | 19.2 (26.8)
  IL-8 pre-dose | 8.7 (2.7) | 2.2 (1.0) | 8.1 (4.7) | 4.0 (2.2) | 11.9 (16.3) | 18.6 (14.7)
  IL-8 4 hour post-dose | 8.2 (3.1) | 2.3 (1.2) | 57.1 (64.0) | 89.8 (144.5) | 10.4 (11.4) | 13.2 (11.1)
  IL-8 24 hour post-dose | 9.0 (2.8) | 5.9 (3.9) | 16.7 (8.2) | 9.8 (1.5) | 25.8 (37.2) | 26.1 (11.2)
  IL-IRA pre-dose | 10.2 (7.7) | 26.4 (26.3) | 29.5 (16.1) | 2.8 (2.1) | 26.5 (42.7) | 1.6 (0)
  IL-IRA 4 hour post-dose | 4.1 (4.3) | 3.3 (2.9) | 1268.5 (1733.8) | 3055.1 (5286.2) | 5.4 (8.6) | 1.6 (0)
  IL-IRA 24 hour post-dose | 5.3 (6.4) | 13.3 (10.2) | 40.5 (8.6) | 4.5 (5.1) | 9.0 (16.6) | 1.6 (0)
  MCP-1 pre-dose | 101.2 (13.1) | 76.5 (59.8) | 70.5 (17.5) | 111.7 (3.52) | 244.5 (210.5) | 164.4 (134.1)
  MCP-1 4 hour post-dose | 90.0 (18.8) | 46.0 (23.6) | 718.8 (872.8) | 1202.5 (1811.4) | 160.2 (117.7) | 137.2 (33.1)
  MCP-1 24 hour post-dose | 162.1 (69.8) | 119.5 (69.0) | 206.9 (118.6) | 184.6 (22.7) | 316.6 (198.4) | 445.8 (337.8)

6. Secondary Outcome: DCR-MYC Biological Activities (Phase 1b Only)
Description: Tumor biopsies (2 total) to be performed in Phase 1b MTD expansion cohort only (6 patients). Patients will have biopsies performed prior to Cycle 1/Day 1 and on Cycle 2/Day 11.
Time Frame: Cycle 1 and 2
Population: Planned expansion into the MTD biopsy cohort and phase 2 portion of the study did not occur due to the sponsor's decision to prematurely end the study.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Tmax (Hr) - DCR-MYC Levels in Blood (Phase 1b Only): Dosing Day 1 and Day 8
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3
hr
  Tmax: Day 1 | 2.4 (0.14) | 2.7 (0.68) | 2.6 (0.27) | 2.9 (0.55) | 2.3 (0.26) | 2.2 (0.14)
  Tmax: Day 8 | 2.6 (0.60) | 2.4 (0.13) | 2.7 (0.35) | 2.2 (0.24) | 3.0 (0.72) | 2.2 (0.24)

8. Secondary Outcome: Cmax_D (kg*ng/mL/mg) - DCR-MYC Levels in Blood (Phase 1b Only): Dosing Day 1 and Day 8
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg*ng/mL/mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 33 | 6 | 3
kg*ng/mL/mg
  Cmax_D: Day 1 | 16832 (10192) | 23952 (17701) | 20652 (2482.5) | 21794 (9098.8) | 28527 (12076) | 23384 (4241.4)
  Cmax_D: Day 8 | 14045 (475.74) | 27525 (16827) | 22095 (3852.7) | 29964 (5724.8) | 30457 (20247) | 31931 (10677)

9. Secondary Outcome: AUClast_D (hr*kg*ng/mL/mg) - DCR-MYC Levels in Blood (Phase 1b Only): Dosing Day 1 and Day 8
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*kg*ng/mL/mg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3
hr*kg*ng/mL/mg
  AUClast_D: Day 1 | 178997 (125460) | 299295 (312426) | 197244 (116908) | 195133 (56544) | 290201 (169069) | 201529 (45290)
  AUClast_D: Day 8 | 163478 (109924) | 739203 (698459) | 389653 (293467) | 350625 (132910) | 274941 (168548) | 383537 (84286)

10. Secondary Outcome: AUClast (hr*ng/mL) - DCR-MYC Levels in Blood (Phase 1b Only): Dosing Day 1 and Day 8
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3
hr*ng/mL
  AUClast : Day 1 | 22375 (15683) | 59859 (62485) | 59173 (35072) | 87810 (25445) | 197337 (114967) | 171299 (38496)
  AUClast : Day 8 | 20435 (13741) | 147841 (139692) | 116896 (88040) | 157781 (59810) | 186960 (114612) | 326006 (71643)

ADVERSE EVENTS:
Time Frame: Throughout entire duration of the study (e.g., approximately 3 month period)
Groups:
- Cohort 1: N = 3, received two, 2-hour infusions of 0.125 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined 5 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 2: N = 3, received two, 2-hour infusions of 0.2 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined 5 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 3: N = 3, received two, 2-hour infusions of 0.3 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined 5 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 4: N = 3, received two, 2-hour infusions of 0.45 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined 5 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 5: N = 6, received two, 2-hour infusions of 0.68 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined 5 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
- Cohort 6: N = 3, received two, 2-hour infusions of 0.85 mg/kg DCR-MYC, once on Day 1 and once on Day 8 within a 21-day cycle. The protocol outlined 5 21-day cycles, each with dosing on days 1 and 8. The study was terminated prematurely and subjects were not treated after the termination date.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/3 | 3/3 | 1/3 | 3/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/3 | 2/6 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=3) | Cohort 5 (N=6) | Cohort 6 (N=3)
Spinal cord compression/ Spinal Cord Compression Due To Pathologic Fracture Of T1 (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain/ Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea/ Increased Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness/ Flu Like Symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome/ Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis/ Cholangitis Due To Pd (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone/ Osteolytic Jaw Lesion Due To Progression Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock/ Hypovolemic Hypoperfusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=3) | Cohort 5 (N=6) | Cohort 6 (N=3)
Fatigue (General disorders) | 0 | 1 | 2 | 2 | 1 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 2 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Influenza-like illness (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
AST increased (Investigations) | 1 | 0 | 2 | 1 | 1 | 1
ALT increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
GGT increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued by the Sponsor because of evolving data from a separate study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR agrees that the Principal Investigator shall have the right to publish or permit the publication of any information or material relating to or arising out of the work after prior submittal to SPONSOR provided that if SPONSOR shall so request, the investigator will delay publication for a maximum of ninety (90) days after submittal to SPONSOR to enable SPONSOR to protect its rights. SPONSOR will comment on such documents within thirty (30) days.